CLINICAL TRIAL: NCT06530446
Title: EFFECT OF SMART PHONE ADDICTION ON ELBOW JOINT PREFORMANCE AMONG ADULTS
Brief Title: SMART PHONE ADDICTION AND ELBOW JOINT PERFORMANCE
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samaa Ahmed Hamed, Researcher Physiotherapist, Cairo University
Other Study IDs: P.T.REC/012/005420
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Elbow Joint Performance, Ms Strength, Proprioception and Elbow Functional Abilities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group: observational study of this group
  Interventions: Other: one group. observational study

INTERVENTIONS:
Other: one group. observational study — observational study of this group

SUMMARY:
smart phone addiction negatively impacted the pain in the muscles of the neck, shoulder, elbow, and the hand. the negative impact of prolonged smartphone use has shown an association between smartphone addiction and musculoskeletal pain in different areas of the body. Caution should be taken towards the safe implementation of smartphone use.

The combination of repetitive movements, poor posture, and over-use of mobile phones for texting or playing games, without taking rest breaks, can cause injury to the nerves, muscles, and tendons in the fingers, hands, wrists, arms, elbows, shoulders, and neck, which if ignored, may lead to long-term damage. Staying stationary for hours with the same hand and elbow movements while using mobile phones not only disrupts the posture of the individual but also causes inefficiency at work. Thus, their prolonged use significantly affects the quality of life as well as the activities of daily life of the individual .No previous study has investigated the link between smartphone addiction and elbow joint performance, to the authors' knowledge. Therefore, the primary purpose of this study will be to determine the relationship between smartphone addiction and elbow joint performance.

ELIGIBILITY:
Inclusion Criteria:

* This study will comprise healthy volunteers between the ages of 18 and 30 who needed to use a smart phone.
* Dominant side will be involved.
* Subjects who put in more than 4 hours per day using smartphone.
* willing to give consent to participate in this study.

Exclusion Criteria:

* recent fracture in neck and upper limb
* any traumatic injury to neck and upper limb prior 6 months
* congenital abnormalities and severe surgical and neurological disorders.
* Pregnant females

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: both female and male, aged between 18- 30 years old
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
MS strength | 6 months
  Hand-held dynamometer (Lafayette )

IPD SHARING:
Plan to Share IPD: Undecided